CLINICAL TRIAL: NCT03892863
Title: A Pilot Study of Repetitive Transcranial Magnetic Stimulation for Improvement of Depression in Amyotrophic Lateral Sclerosis
Brief Title: Repetitive Transcranial Magnetic Stimulation as Therapy for Depression in Amyotrophic Lateral Sclerosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Participants were not able to stay for two weeks near our center.
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Jakub Antczak, Principal Investigator, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JagiellonianU61
Record Dates: First submitted 2019-03-26; First posted 2019-03-27 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; depression; rTMS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Depression

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to real or placebo (sham) stimulation.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Sham stimulation will be provided by holding the stimulating coil perpendicularly to the scalp, which assures similar impression as during active stimulation but prevents significant magnetic field to reach the brain tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active repetitive transcranial magnetic stimulation (Active Comparator): 10 hertz (Hz) rTMS will be administered over the left dorsolateral prefrontal cortex. Therapy will include 10 daily sessions (on consecutive week days). In every sessions 3000 magnetic pulses of 120% of the resting motor threshold intensity will be elicited.
  Interventions: Device: active repetitive transcranial magnetic stimulation
- sham repetitive transcranial magnetic stimulation (Sham Comparator): Sham stimulation will mimic the active one except that the stimulating coil will be held perpendicularly to the scalp, which assures similar impression as the active stimulation but prevents that significant magnetic field will reach brain tissue.
  Interventions: Device: sham repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: active repetitive transcranial magnetic stimulation — High frequency rTMS to induce the long term potentiation in the left dorsolateral prefrontal cortex
  Arms: active repetitive transcranial magnetic stimulation
Device: sham repetitive transcranial magnetic stimulation — High frequency rTMS to induce the long term potentiation in the left dorsolateral prefrontal cortex
  Arms: sham repetitive transcranial magnetic stimulation

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a neurodegenerative disease characterized by progressive loss of central and peripheral motor neurons. ALS leads to death usually within 3 to 5 years from the onset of the symptoms. Available treatment can prolong the disease duration but cannot modify the disease course. Depression is a frequent complication of ALS, which further decreases quality of life and the available data concerning effectivity of antidepressant drugs are conflicting. Repetitive Transcranial Magnetic Stimulation (rTMS) is a noninvasive method of modulation of brain plasticity with confirmed antidepressive effect. The purpose of this study is to compare the effectiveness of rTMS in improving the depression in patients with ALS with placebo stimulation. Intervention will include 10 daily sessions. In each session 3000 magnetic pulses will be administered over the left dorsolateral prefrontal cortex. Assessment depression severity will be made before and after therapy, as well as two and four weeks later.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a neurodegenerative disease characterized by progressive loss of central and peripheral motor neurons. ALS leads to death usually within 3 to 5 years from the onset of the symptoms. Available treatment can prolong the disease duration but cannot modify the disease course. Depression is a frequent complication of ALS, which further decreases quality of life and the available data concerning effectivity of antidepressant drugs are conflicting. Similarly, the apathy may also complicate ALS and worsen the prognosis. Repetitive Transcranial Magnetic Stimulation (rTMS) is a noninvasive method of modulation of brain plasticity with proved antidepressive effect in patients suffering from major depression and in depression associated with several neurological disorders such as Parkinson's disease or stroke.

The purpose of this study is to compare the effectiveness rTMS in improving the depression and - as a secondary outcome - the apathy and daily functioning in patients with ALS.

Intervention will include ten daily sessions of rTMS. In each session 3000 magnetic pulses will be administered over the left dorsolateral prefrontal cortex. Stimulation intensity will equal 120% of the motor threshold value for the right first dorsal interosseus.

Assessment of depression severity and of apathy and daily functioning will be made before and after therapy, as well as two and four weeks later.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of definite or probable ALS according to el Escorial criteria (Brooks et al. 2000)
* Depression defined as the score in Beck's Depression Inventory ≥14
* Mini-Mental State Examination score ≥26

Exclusion Criteria:

* Psychiatric symptoms, which may negatively influence patient's tolerance and adherence to therapy
* Respiratory insufficiency and other complications od advanced stages of ALS, which may compromise patient's ability to undergo the study procedure
* Contraindications for rTMS as listed by the Guidelines of the International Federation of Clinical Neurophysiology (Rossi et al. 2009) i.e. seizure in the past, epilepsy, presence of magnetic material in the reach of magnetic field, pregnancy, likelihood to get pregnant, intracranial electrodes, cardiac pacemaker or intracardiac lines, frequent syncopes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-15 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Beck's Depression Inventory ater rTMS, total score, range 0 to 63, with higher values representing a worse outcome | Before rTMS, directly (on the same day) after finishing rTMS
  Change from baseline score in the Beck's Depression Inventory to the measurement taken directly after finishing rTMS.
Beck's Depression Inventory first follow up, total score, range 0 to 63, with higher values representing a worse outcome | Before rTMS, two weeks after finishing rTMS
  Change from baseline score in the Beck's Depression Inventory to the measurement taken two weeks after finishing rTMS.
Beck's Depression Inventory second follow up, total score, range 0 to 63, with higher values representing a worse outcome | Before rTMS, four weeks after finishing rTMS
  Change from baseline score in the Beck's Depression Inventory to the measurement taken four weeks after finishing rTMS.

SECONDARY OUTCOMES:
Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised after rTMS, total score, range 0 to 40 with higher values representing a better outcome | Before rTMS, directly (on the same day) after finishing rTMS
  Change from baseline score in the Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised to the measurement taken directly after finishing rTMS.
Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised first follow up, total score, range 0 to 40 with higher values representing a better outcome | Before rTMS, two weeks after finishing rTMS
  Change from baseline score in the Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised to the measurement taken two weeks after finishing rTMS.
Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised second follow up, total score, range 0 to 40 with higher values representing a better outcome | Before rTMS, four weeks after finishing rTMS
  Change from baseline score in the Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised to the measurement taken directly after finishing rTMS.
Apathy Evaluation Scale Clinical Version ater rTMS, total score, range 18 to 72 with higher values representing a worse outcome | Before rTMS, directly (on the same day) after finishing rTMS
  Change from baseline score in the Apathy Evaluation Scale Clinical Version to the measurement taken taken directly after finishing rTMS.
Apathy Evaluation Scale Clinical Version first follow up, total score, range 18 to 72 with higher values representing a worse outcome | Before rTMS, two weeks after finishing rTMS
  Change from baseline score in the Apathy Evaluation Scale Clinical Version to the measurement taken two weeks after finishing rTMS.
AES-C second follow up, total score, range 18 to 72 with higher values representing a worse outcome | Before rTMS, four weeks after finishing rTMS
  Change from baseline score in the Apathy Evaluation Scale Clinical Version to the measurement taken four weeks after finishing rTMS.

CONTACTS AND LOCATIONS:
Overall Officials: Jakub M Antczak, MD, Principal Investigator — Department of Neurology, Jagiellonian University Medical College
Locations (1):
- Jagiellonian University Medical College, Department of Neurology, Krakow, Poland

IPD SHARING:
Plan to Share IPD: Yes
After completing the study, the details of neurophysiologic diagnostics including motor threshold, the age and gender as well as individual scores of Mini-Mental State Examination, Beck depression inventory, AES-C and Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised will be made available to other researchers on request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available after the study is published.
Access Criteria: On request send by e-mail: jantczak@cm-uj.krakow.pl

REFERENCES:
- [Background] Brooks BR, Miller RG, Swash M, Munsat TL; World Federation of Neurology Research Group on Motor Neuron Diseases. El Escorial revisited: revised criteria for the diagnosis of amyotrophic lateral sclerosis. Amyotroph Lateral Scler Other Motor Neuron Disord. 2000 Dec;1(5):293-9. doi: 10.1080/146608200300079536. No abstract available. PMID 11464847
- [Background] Fregni F, Santos CM, Myczkowski ML, Rigolino R, Gallucci-Neto J, Barbosa ER, Valente KD, Pascual-Leone A, Marcolin MA. Repetitive transcranial magnetic stimulation is as effective as fluoxetine in the treatment of depression in patients with Parkinson's disease. J Neurol Neurosurg Psychiatry. 2004 Aug;75(8):1171-4. doi: 10.1136/jnnp.2003.027060. PMID 15258224
- [Background] Lefaucheur JP, Andre-Obadia N, Antal A, Ayache SS, Baeken C, Benninger DH, Cantello RM, Cincotta M, de Carvalho M, De Ridder D, Devanne H, Di Lazzaro V, Filipovic SR, Hummel FC, Jaaskelainen SK, Kimiskidis VK, Koch G, Langguth B, Nyffeler T, Oliviero A, Padberg F, Poulet E, Rossi S, Rossini PM, Rothwell JC, Schonfeldt-Lecuona C, Siebner HR, Slotema CW, Stagg CJ, Valls-Sole J, Ziemann U, Paulus W, Garcia-Larrea L. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS). Clin Neurophysiol. 2014 Nov;125(11):2150-2206. doi: 10.1016/j.clinph.2014.05.021. Epub 2014 Jun 5. PMID 25034472
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Shen X, Liu M, Cheng Y, Jia C, Pan X, Gou Q, Liu X, Cao H, Zhang L. Repetitive transcranial magnetic stimulation for the treatment of post-stroke depression: A systematic review and meta-analysis of randomized controlled clinical trials. J Affect Disord. 2017 Mar 15;211:65-74. doi: 10.1016/j.jad.2016.12.058. Epub 2017 Jan 10. PMID 28092847